CLINICAL TRIAL: NCT03181191
Title: The Anatomical Location, Cellular Origin and Molecular Basis of Gut-derived Glucagon Secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Consultant endocrinologist, Professor of Clinical Endocrinology and Director of Center for Clinical Metabolic Research, University Hospital, Gentofte, Copenhagen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UHG-CFD-PX-BIOPSY
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Totally pancreatectomised patients (Active Comparator): Oral glucose tolerance test and biopsies
  Interventions: Other: Oral glucose tolerance test
- Type 2 diabetes patients (Active Comparator): Oral glucose tolerance test and biopsies
  Interventions: Other: Oral glucose tolerance test
- Healthy control subjects (Active Comparator): Oral glucose tolerance test and biopsies
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — Oral glucose tolerance test and biopsies

SUMMARY:
Delineation of the anatomical location, cellular origin and molecular basis of gut-derived glucagon secretion

DETAILED DESCRIPTION:
Aim: to delineate the anatomical origin, the molecular structure and precursors, the regulation and the (patho-) physiological implications of gut-derived glucagon.

Eight totally pancreatectomised patients, eight type 2 diabetes patients and eight healthy controls (age 18-80, BMI <30) with normal kidney and liver parameters and hgb> 6.5 - will be included. The participants will each undergo one screening day and one study day including a gastroduodenoscopy. Multiple biopsies will be taken at several predefined locations in the upper gastrointestinal tract. These biopsies will be analysed with different techniques including immunohistochemical staining, quantitative polymerase chain reaction (qPCR-) analyses and more to search for glucagon. After the last biopsy has been collected, 50 g of glucose dissolved in 100 ml water is infused through the enteroscope into the most proximal part of the small intestine. Hereafter blood samples for glucagon and gut hormone analyses will be collected 15, 30 and 45 min after the glucose infusion.

ELIGIBILITY:
Inclusion Criteria:

* normal kidney function, normal liver function, normal hemoglobin levels

Exclusion Criteria:

* diabetes type 1, first degree relatives with type 2 diabetes

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2017-12-03 (Actual); Study Completion 2017-12-03 (Actual)

PRIMARY OUTCOMES:
gut-derived glucagon | 1 year
  The primary objective is to investigate mucosal biopsies from specific regions of the upper gastrointestinal tract

SECONDARY OUTCOMES:
Oral glucose tolerance test | 45 minutes
  Glucose metabolism - hormones, insulin, glucagon, glp-1

CONTACTS AND LOCATIONS:
Overall Officials: Filip Knop, MD, PhD, Study Director — University Hospital, Gentofte, Copenhagen
Locations (1):
- Center for Diabetes Research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: No